CLINICAL TRIAL: NCT00407979
Title: Analysis and Correlation of Cathelicidin Expression in Skin and Saliva of Subjects With Atopic Dermatitis and Psoriasis
Brief Title: Comparison of Cathelicidin Expression in Skin and Saliva in Patients With Atopic Dermatitis and Psoriasis
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT ADVN CATH 02; DAIT-ADVN-CATH-02
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Atopic Dermatitis; Psoriasis
MeSH Terms: conditions — Dermatitis, Atopic; Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, skin, and saliva samples will be retained

GROUPS / COHORTS (4):
- People with Atopic Dermatitis
- People with Psoriasis
- Generally healthy people
- People with Atopic Dermatitis and Eczema Herpeticum

SUMMARY:
Cathelicidins are small proteins in the human body that protect against infection. The purpose of this study is to determine if the amount of cathelicidins and other small proteins found in saliva can predict the amount of these in the skin of people who have acute atopic dermatitis (AD) or psoriasis.

DETAILED DESCRIPTION:
People with AD or psoriasis are very sensitive to skin infections and inflammations. A group of small proteins known as cathelicidins are known to be responsible for immune defense against such infections. People with AD or psoriasis seem to be missing these proteins from their skin. The purpose of this study is to determine if the amount of cathelicidins and other small proteins in saliva is a predictor for the amount found in the skin.

This is a single visit observational study. People with AD or psoriasis, as well as healthy participants, are being recruited for this study. Participants will provide a detailed medical history and undergo a physical examination. In addition, saliva and blood collection, and skin punch biopsies will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of typical AD for at least 6 months as defined by ADVN standardized diagnostic criteria OR diagnosis of typical plaque psoriasis for at least 6 months
* ADEH participants as defined by ADVN standardized diagnostic criteria
* Healthy participants with no personal or family history of food allergy, AD, asthma, or allergic rhinitis
* Persons residing in the US
* Healthy individuals with no systemic disorders as outlined in the exclusion criteria
* Subjects 18 to 70 years of age
* Male or female

Exclusion Criteria for All Participants:

* Under 18 or over 70 years of age
* Presence of allergic hypersensitivity without stringent AD features, allowing only a presumptive diagnosis of AD
* Presence of AD with exfoliative erythroderma
* Presence of psoriasis with exfoliative erythroderma or presence of guttate psoriasis, primary palmoplantar psoriasis, or pustular psoriasis
* Ongoing dental disease (e.g., gingivitis)
* Bleeding disorder
* Presence of AD or psoriasis in which temporarily stopping current medications would cause worsening of the disease (Participants with active ADEH will be allowed to continue medication)
* Systemic immunosuppressive or chemotherapeutic agents, anti-inflammatory biologics (e.g., alefacept, etanercept), or oral calcineurin inhibitors within 30 days of screening visit
* Topical corticosteroids, oral or topical antibiotics, oral antivirals, immune enhancers (e.g., imiquimod), or topical calcineurin inhibitors within 7 days prior to screening visit (Participants with active ADEH will be allowed to continue medication)
* Receiving phototherapy (e.g., ultraviolet light B [UVB], psoralen plus ultraviolet light A [PUVA]) within 30 days of study entry
* Autoimmune disease or immunodeficiency
* Active fungal, bacterial, or viral infections (Except ADEH subjects)
* Active systemic cancer. Participants with uncomplicated nonmelanoma skin cancer are not excluded.
* Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the study
* Diabetic requiring medication
* Pregnancy or breastfeeding
* Inability or unwillingness of a participant to give written informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Generally healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2005-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To measure the local and systemic expression of cathelicidin (hCAP18/LL-37) in subjects with ADEH-, ADEH+, psoriasis, and in normal controls. | 18 months

SECONDARY OUTCOMES:
To determine whether the relative abundance of cathelicidins (hCAP18/LL-37) in the skin correlates with the expression in saliva and/or blood. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gallo, MD, PhD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - University of California, San Diego, San Diego, California
  - National Jewish Health, Denver, Colorado

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Background] Tomasinsig L, Zanetti M. The cathelicidins--structure, function and evolution. Curr Protein Pept Sci. 2005 Feb;6(1):23-34. doi: 10.2174/1389203053027520. PMID 15638766
- [Result] Schauber J, Dorschner RA, Yamasaki K, Brouha B, Gallo RL. Control of the innate epithelial antimicrobial response is cell-type specific and dependent on relevant microenvironmental stimuli. Immunology. 2006 Aug;118(4):509-19. doi: 10.1111/j.1365-2567.2006.02399.x. PMID 16895558
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY5 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY5 — ImmPort study identifier is SDY5
- Available data/document: Study design, -schedule of events, -demographics, -adverse events, -interventions, -files: SDY5 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY5 — ImmPort study identifier is SDY5